CLINICAL TRIAL: NCT04244383
Title: Expression of Inflammasomes in HCV Patients Before and After Treatment
Brief Title: Expression of Inflammasomes in HCV Patients
Acronym: Inflammasome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Fergany, princible inverstigator, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: ِAssiutU
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: chronic hepatitis C virus patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic hepatitis C virus patients (Experimental): 50 chronic hepatitis C virus patients taking will be trated with direct acting antiviral treatment with three months regimen (Sofosbuvir + Daclatasvir).
  Interventions: Diagnostic Test: interleukin IL-1beta and interleukin IL-18
- treated chronic hepatitis C virus patients (Experimental): the selected 50 chronic hepatitis C virus patients received direct acting antivirals: Sofosbuvir 400 mg and Daclatasvir 60 mg daily for 12 weeks and were assessed for sustained virological response at 12 weeks following the end of treatment (SVR12).
  Interventions: Diagnostic Test: interleukin IL-1beta and interleukin IL-18

INTERVENTIONS:
Diagnostic Test: interleukin IL-1beta and interleukin IL-18 — pro-inflammatory cytokines measured in the serum

SUMMARY:
Hepatitis C virus has been identified a quarter of a decade ago as a leading cause of chronic viral hepatitis that can lead to cirrhosis and hepatocellular carcinoma. Only a minority of patients can clear the virus spontaneously during acute infection. Elimination of HCV during acute infection correlates with a rapid induction of innate and a delayed induction of adaptive immune responses. The majority of patients is unable to clear the virus and develops viral persistence despite the ongoing innate and adaptive immune response. The virus usually develops several strategies to escape these immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C virus patients.
* Patients do not start treatment protocol.

Exclusion Criteria:

* Pregnant women.
* Hepato-cellular carcinoma patients.
* Autoimmune disease patients.
* Patients with liver cirrhosis.
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
changes in the exprssion level of inflammasomes | 6 monthes
  observe the changes in the exprssion level of inflammasomes in the selected chronic HCV patients before treatment with Sofosbuvir 400 mg and Daclatasvir 60 mg daily for 12 weeks and after sustained virological response at 12 weeks following the end of treatment (SVR12).

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Salah El-dien Gaber, lecturer, Principal Investigator — participator in the research; Mohamed Ahmed Medhat, lecturer, Principal Investigator — participator in the research; Sara Fergany Abd El-hamid, student, Principal Investigator — participator in the research

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen H, He G, Chen Y, Zhang X, Wu S. Differential Activation of NLRP3, AIM2, and IFI16 Inflammasomes in Humans with Acute and Chronic Hepatitis B. Viral Immunol. 2018 Nov;31(9):639-645. doi: 10.1089/vim.2018.0058. Epub 2018 Sep 15. PMID 30222506
- [Background] Kanneganti TD. Central roles of NLRs and inflammasomes in viral infection. Nat Rev Immunol. 2010 Oct;10(10):688-98. doi: 10.1038/nri2851. Epub 2010 Sep 17. PMID 20847744
- [Background] YingLi H, Shumei L, Qian Y, Tianyan C, Yingren Z, Wei C. Proapoptotic IL-18 in patients with chronic hepatitis C treated with pegylated interferon-alpha. Clin Exp Med. 2009 Jun;9(2):173-8. doi: 10.1007/s10238-009-0041-5. Epub 2009 Feb 24. PMID 19238512
- [Background] Burchill MA, Roby JA, Crochet N, Wind-Rotolo M, Stone AE, Edwards MG, Dran RJ, Kriss MS, Gale M Jr, Rosen HR. Rapid reversal of innate immune dysregulation in blood of patients and livers of humanized mice with HCV following DAA therapy. PLoS One. 2017 Oct 17;12(10):e0186213. doi: 10.1371/journal.pone.0186213. eCollection 2017. PMID 29040318
- [Background] Shi J, Li Y, Chang W, Zhang X, Wang FS. Current progress in host innate and adaptive immunity against hepatitis C virus infection. Hepatol Int. 2017 Jul;11(4):374-383. doi: 10.1007/s12072-017-9805-2. Epub 2017 Jun 22. PMID 28643186